CLINICAL TRIAL: NCT02252367
Title: Double-blind, Placebo-controlled Study on Men With Lower Urinary Tract Symptoms to Assess Changes in Pressure Flow Study and in Molecular Profile of Prostatic Tissue After 12 Weeks Treatment With Tadalafil.
Brief Title: Effect of 12 Weeks Treatment With Tadalafil vs Placebo on Lower Urinary Tract Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florence (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Mario Maggi, Full Professor of Endocrinology, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANDRO-AOUC-2014-01
Record Dates: First submitted 2014-09-22; First posted 2014-09-30 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Phosphodiesterase 5 Inhibitors; BPH/LUTS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental): 43 male subjects affected by BPH (benign prostatic hyperplasia) planned for simple prostatectomy will be randomized to tadalafil 5 mg - 1 film-coated tablet orally once daily for 12 weeks.
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): 43 male subjects affected by BPH (benign prostatic hyperplasia) planned for simple prostatectomy will be randomized to placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil 5 mg once daily for 12 weeks.
  Other Names: Cialis
  Arms: Tadalafil
Other: Placebo — Placebo tablet once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
At present time several preclinical and clinical study have demonstrated the safety and efficacy of PDE5 (phosphodiesterase type 5)-inhibitors for LUTS/BPH (lower urinary tract symptoms/benign prostatic hyperplasia) patients with or without erectile dysfunction. However, the link between clinical outcomes (symptoms scores), functional activity (urodynamic findings) and molecular pathways, in particular regarding inflammatory pattern (molecular analyses), has not been previously investigated.

Aim of present study is to assess, for the first time in literature, changes in pressure flow study (PFS) and changes in molecular profile of prostatic tissue (inflammatory and tissue remodeling markers) in men treated for 12 weeks with tadalafil 5 mg compared with placebo and to correlate these data with changes in symptoms scores (IPSS, International Prostatic Symptoms Score) in men with LUTS secondary to BPH refractory to alpha blockers.

ELIGIBILITY:
Inclusion Criteria:

* adult male subjects planned to undergo simple prostatectomy (TURP, Transurethral resection of the prostate, or open prostatectomy) for benign prostatic hyperplasia;
* treatment with alpha-blockers (Tamsulosin 0.4 mg/die)
* being capable of giving informed consent.

Exclusion Criteria:

* participation in another clinical study;
* known or suspected presence of prostatic cancer or PSA (prostate specific antigen) value >10 ng/mL;
* suspected lack of the participant's compliance;
* known severe allergies or hypersensitivity to the study drug (active substance or excipients of the formulation);
* nown neurogenic bladder (i.e. Parkinson's disease);
* suspected or proven urinary infections;
* presence of bladder stone.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Improvement of LUTS/BPH symptoms | 12 weeks
  BPH-associated inflammatory symptoms will be assessed by using the National Institute of Health Chronic Prostatitis Symptom Index (NIH-CPSI). BPH-associated LUTS will be assessed by using International Prostate Symptom Score (IPSS).

SECONDARY OUTCOMES:
Improvement of pressure flow study (PFS) parameters | 12 weeks
  Maximum flow rate (Qmax), average flow rate (Qave), voided volume (Vcomp), post void residual volume (PVR) will be evaluated. An abdominal ultrasound immediately after voiding for uroflowmetry will be performed in order to determine the PVR.
Volumetric change of the prostate | 12 weeks
  Prostate volume as assessed by transrectal ultrasound
Change in prostate inhomogeneity and in the number of prostatic macrocalcifications | 12 weeks
  BPH-associated prostate inhomogeneity and presence of micro-calcifications will be assessed by using male genital tract male genital tract colour-Doppler ultrasonography.
Variation in genic expression of prostatic inflammation markers | 12 weeks
  BPH-associated prostate inflammation, fibrosis, and hypoxia will be measured by immunohistochemical and quantitative RT-PCR (qRT-PCR) analyses of inflammatory-, fibrosis- and hypoxia-related markers.
Variation in serum inflammation markers CRP (C-reactive protein) and ESR (Erythrocyte Sedimentation Rate) | 12 weeks
  CRP measured on serum and ESR measured on blood drawn at baseline and after 12 weeks
Improvement in metabolic profile | 12 weeks
  Metabolic parameters will be evaluated (glycaemia, insulinemia, total cholesterol, HDL, triglycerides, HbA1c, mean arterial pressure, waist circumference, body mass index)
Variation in seminal plasma IL-8 (interleukin-8) levels | 12 weeks
  Seminal IL-8, a chemokine involved in male genital tract infection/inflammation, will be evaluated.
Improvement in erectile function | 12 weeks
  Erectile function will be assessed by using the International Index of Erectile Function-5 (IIEF-5) score.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maggi, Principal Investigator — University of Florence
Locations (1):
- Clinica Urologica - Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

REFERENCES:
- [Background] Gacci M, Corona G, Salvi M, Vignozzi L, McVary KT, Kaplan SA, Roehrborn CG, Serni S, Mirone V, Carini M, Maggi M. A systematic review and meta-analysis on the use of phosphodiesterase 5 inhibitors alone or in combination with alpha-blockers for lower urinary tract symptoms due to benign prostatic hyperplasia. Eur Urol. 2012 May;61(5):994-1003. doi: 10.1016/j.eururo.2012.02.033. Epub 2012 Feb 25. PMID 22405510
- [Background] Gacci M, Vittori G, Tosi N, Siena G, Rossetti MA, Lapini A, Vignozzi L, Serni S, Maggi M, Carini M. A randomized, placebo-controlled study to assess safety and efficacy of vardenafil 10 mg and tamsulosin 0.4 mg vs. tamsulosin 0.4 mg alone in the treatment of lower urinary tract symptoms secondary to benign prostatic hyperplasia. J Sex Med. 2012 Jun;9(6):1624-33. doi: 10.1111/j.1743-6109.2012.02718.x. Epub 2012 Apr 17. PMID 22510238